CLINICAL TRIAL: NCT01402219
Title: Nephrotoxicity of Iopamidol Versus Iodixanol in High-Risk Patients:A Multicentre Randomized Double-Blind Trail of Contrast-Induced Nephropathy in Patients With Chronic Kidney Disease
Brief Title: Nephrotoxicity of Iopamidol Versus Iodixanol in High-Risk Patients
Acronym: NEIHR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There were few eligible subjects from other centers.
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, Jiyan Chen, MD, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2008A030201002
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Renal Disease
Keywords: contrast-induced nephropathy; contrast medium; creatinine clearance; coronary angiography; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — iodixanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Iopamiro-370 (Active Comparator)
  Interventions: Drug: Iopamidol injection 76%
- Visipaque 320 (Active Comparator)
  Interventions: Drug: iodixanol

INTERVENTIONS:
Drug: Iopamidol injection 76% — Iopamiro-370 (Iopamidol injection 76%) is provided in single dose bottles/vials, ready to use, aqueous, nonpyrogenic, colorless to pale yellow sterile solution
  Arms: Iopamiro-370
Drug: iodixanol — Visipaque 320 (iodixanol) injection is provided in bottles/flexible containers, ready to use sterile, pyrogen-free colorless to pale yellow solution
  Arms: Visipaque 320

SUMMARY:
The purpose of this study is to compare the incidence of contrast-induced nephropathy (CIN) following the administration of iopamidol-370 (Iopamiro-370) and iodixanol-320 (Visipaque 320) in patients with chronic kidney disease undergoing coronary angiography.

DETAILED DESCRIPTION:
To compare the incidence of contrast-induced nephropathy (CIN)(an absolute SCr increase 0.5 mg/dL from baseline) following the administration of iopamidol-370 (Iopamiro-370) and iodixanol-320 (Visipaque 320) in patients with chronic kidney disease (serum creatinine level more than 1.5 mg/dL for men and more than 1.3 mg/dL for women or preprocedural estimated glomerular ﬁltration rate(eGFR):15-60 mL/min/1.73 m2) undergoing coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* Provides written Informed Consent and is willing to comply with protocol requirements
* Is ≥18 years of age
* Has a documented predose serum creatinine level of ≥1.5 mg/dL for men and ≥ 1.3 mg/dL for women or predose estimated glomerular ﬁltration rate (eGFR) of > 15 and ≤ 60 mL/min/1.73 m2, calculated via the MDRD formula from a SCr obtained within 72 hours of enrollment into the study;
* Is referred for cardiac angiography with or without PCI;
* If at the discretion of the Investigator is receiving or will be receiving a prophylactic medication for renal function, the medication is one that is permitted by this protocol (N acetylcysteine, 1200 mg twice daily on the day before and on the day of the cardiac angiography procedure);
* Undergoes or is scheduled to undergo pre, peri, or post procedure hydration permitted by this protocol, i.e.:
* 154 mEq/L sodium bicarbonate solution, administered intravenously at 3 mL/kg/hr for 1 hour before cardiac angiography, followed by an infusion of 1 mL/kg/hr during and out to 6 hours after cardiac angiography, or 0.9% normal saline administered intravenously at 1 mL/kg/hr for 8-12 hours before cardiac angiography, followed by an infusion of 1 mL/kg/hr during and out to 24 hours after cardiac angiography,for the patients with left ventricular ejection fraction <35% or congestive heart failure (class III in accordance with the classification of the New York Heart Association (NYHA), the rate of infusion decreases to half of the above ordinary rate.

Exclusion Criteria:

* Is a pregnant or lactating female. Exclude the possibility of pregnancy: by laboratory testing on-site at the institution (measurement of serum or urine βHCG) within 24 hours prior to the start of investigational product administration by history (e.g., tubal ligation or hysterectomy, post menopausal with a minimum 1 year without menses)
* Has a history of hypersensitivity to iodine-containing compounds;
* Has unstable renal function (i.e., acute worsening of renal function, as determined by the Investigator, that has been observed in the 7 days prior to enrollment) and/or is in acute renal failure;
* Has end-stage renal disease (i.e., eGFR <15 mL/min/1.73 m2)
* Has severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association (NYHA) ;
* Has uncontrolled diabetes, as determined by the Investigator;
* Has received an iodinated contrast agent within 7 days prior to the administration of the study agent or is scheduled to receive an iodinated contrast agent within 72 hours after administration of the study agent; intake of nephrotoxic drugs within the previous seven days Prior to, during or post the cardiac angiography, is receiving or will be receiving a prophylactic medication to prevent acute kidney injury that is not permitted by this protocol (e.g., theophylline, fenoldopam, etc.);
* Is planned to undergo major surgery (e.g. CABG, valve surgery, etc.) within 48-72 hours after contrast administration;
* Is planned to receive an intravenous diuretic or mannitol as prophylaxis to prevent acute renal injury (Note: chronic administration is allowed);
* Is hemodynamically unstable within 48 hours pre-contrast administration defined as a systolic blood pressure < 90 mmHg or requires pressor or intra-aortic balloon support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2008-11; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
contrast-induced nephropathy | 48-72 h
  Contrast-Induced Nephropathy was defined as an increase in serum creatinine of more than 0.5 mg/dl or 25% from the baseline within 48-72 h of contrast exposure

SECONDARY OUTCOMES:
A relative increase in serum creatinine | 48-72 h
  A relative increase in serum creatinine was defined as more than 25% increase in serum creatinine within 48-72 h of contrast exposure.
A relative increase in estimated glomerular ﬁltration rate (eGFR) | 48-72 h
  A relative increase in eGFR was defined as more than 25% increase in eGFR within 48-72 h of contrast exposure
An absolute increase in serum creatinine | 48-72 h
  An absolute increase in serum creatinine within 48-72 h of contrast exposure
Major adverse clinical events | 1 month
  Major adverse clinical events: death, requiring renal replacement therapy, 2nd myocardial infarction,target revascularization,acute heart failure, mechanical ventilation,2nd angina,tachyarrhythmia,hypotension,intra-aortic balloon pump and stroke
Major adverse clinical events | 1 year
  Major adverse clinical events: death, requiring renal replacement therapy, acute myocardial infarction,target revascularization,acute heart failure, mechanical ventilation,2nd angina,tachyarrhythmia,hypotension,intra-aortic balloon pump and stroke
An significant increase in serum creatinine | 48-72 h
  An significant increase in serum creatinine was defined as an increase in serum creatinine of more than 1.0 mg/dl from the baseline within 48-72 h of contrast exposure
Contrast-Induced Acute Kidney Injury | 48 h
  Contrast-Induced Acute Kidney Injury was defined as an increase in serum creatinine concentration of more than 0.3 mg/dL from the baseline value at 48 hours after administration of the contrast exposure or the need for dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, MD, Study Chair — chen-jiyan@163.com; Yingling Zhou, MD, Study Director — Guangdong Cardiovascular Institute,Guangdong General Hospital; Yong Liu, MD, Principal Investigator — liuyongyisheng@126.com
Locations (1):
- Guangdong Cardiovascular Institute,Guangdong General Hospital, Guangzhou, Guangdong, China